CLINICAL TRIAL: NCT01984814
Title: The Effect of Autologous Bone Marrow Mononuclear Cell Transplantation on the Survival Duration in Amyotrophic Lateral Sclerosis - A Retrospective Control Study
Brief Title: Stem Cell Therapy for Amyotrophic Lateral Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-04
Record Dates: First submitted 2013-11-08; First posted 2013-11-15 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem cell (Experimental): Autologous bone marrow mononuclear cells intrathecal and intramuscular transplantation
  Interventions: Biological: Stem cell
- Control (No Intervention): No cell transplantation was done

INTERVENTIONS:
Biological: Stem cell — Autologous bone marrow derived mononuclear cells were administered via intrathecal and intramuscular routes.
  Arms: Stem cell

SUMMARY:
The effect of autologous bone marrow mononuclear cells on duration of survival in Amyotrophic Lateral Sclerosis patients.

DETAILED DESCRIPTION:
Survival duration in Amyotrophic Lateral Sclerosis patients who received cellular transplantation was compared to patients who did not receive cellular transplantation. Kaplan-Meier survival analysis was used for this comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnoses of definite amyotrophic lateral sclerosis.
* Clear information about date of onset of symptoms, documented contact information and follow up information

Exclusion Criteria:

* Patients with diagnoses of Progressive Lateral sclerosis, Progressive bulbar plasy, Progressive spinal muscular atrophy, Progressive muscular atrophy, monomelicamyotrophy or madras motor neuron disease.
* patients with co-morbidities like presence of acute infections such as Human Immunodeficiency Virus/Hepatitis B Virus/Hepatitis C Virus, malignancies, bleeding tendencies, renal failure, severe liver dysfunction and other acute medical conditions such as respiratory infection and pyrexia.

Ages: 26 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Duration of survival | 56 months

CONTACTS AND LOCATIONS:
Overall Officials: Alok K Sharma, MS,MCh, Principal Investigator — Neurogen Brain and Spine Institute
Locations (1):
- Neurogen brain and spine institute, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Chio A, Logroscino G, Traynor BJ, Collins J, Simeone JC, Goldstein LA, White LA. Global epidemiology of amyotrophic lateral sclerosis: a systematic review of the published literature. Neuroepidemiology. 2013;41(2):118-30. doi: 10.1159/000351153. Epub 2013 Jul 11. PMID 23860588
- [Background] Deda H, Inci MC, Kurekci AE, Sav A, Kayihan K, Ozgun E, Ustunsoy GE, Kocabay S. Treatment of amyotrophic lateral sclerosis patients by autologous bone marrow-derived hematopoietic stem cell transplantation: a 1-year follow-up. Cytotherapy. 2009;11(1):18-25. doi: 10.1080/14653240802549470. PMID 19012065
- [Background] Blanquer M, Moraleda JM, Iniesta F, Gomez-Espuch J, Meca-Lallana J, Villaverde R, Perez-Espejo MA, Ruiz-Lopez FJ, Garcia Santos JM, Bleda P, Izura V, Saez M, De Mingo P, Vivancos L, Carles R, Jimenez J, Hernandez J, Guardiola J, Del Rio ST, Antunez C, De la Rosa P, Majado MJ, Sanchez-Salinas A, Lopez J, Martinez-Lage JF, Martinez S. Neurotrophic bone marrow cellular nests prevent spinal motoneuron degeneration in amyotrophic lateral sclerosis patients: a pilot safety study. Stem Cells. 2012 Jun;30(6):1277-85. doi: 10.1002/stem.1080. PMID 22415951
- See also: The Amyotrophic lateral sclerosis association encourages scientific research to find a cure for ALS and heightens awareness of the nature of the disease. — http://www.alsa.org/